CLINICAL TRIAL: NCT05702879
Title: An Early Combined Microbiota and Metabolic Signature in Ulcerative Colitis Patients Predict the Clinical Success of Anti-inflammatory Therapy
Brief Title: Combined Microbiota and Metabolic Signature in Ulcerative Colitis Predicts Anti-Inflammatory Therapy Success
Acronym: COMMIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-02008
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod; Tumor Necrosis Factor Inhibitors; Infliximab; Adalimumab; Etanercept; golimumab; Certolizumab Pegol; Steroids; vedolizumab; Ustekinumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples collected by patients and healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ulcerative colitis patients: Patients with a flare of ulcerative colitis who meet the inclusion criteria. 120 patients will be included.
  Interventions: Drug: Ozanimod; Drug: TNF Inhibitor; Drug: Steroids; Drug: Vedolizumab; Drug: Ustekinumab
- Controls: For each patient, enrollment of a healthy control individual who shares the same living conditions (e.g., spouse or roommate) is attempted

INTERVENTIONS:
Drug: Ozanimod — Start of standard therapy
  Groups: Ulcerative colitis patients
Drug: TNF Inhibitor — Start of standard therapy
  Other Names: infliximab, adalimumab, etanercept, golimumab, and certolizumab.
  Groups: Ulcerative colitis patients
Drug: Steroids — Start of standard therapy
  Other Names: Prednisolon
  Groups: Ulcerative colitis patients
Drug: Vedolizumab — Start of standard therapy
  Groups: Ulcerative colitis patients
Drug: Ustekinumab — Start of standard therapy
  Groups: Ulcerative colitis patients

SUMMARY:
The primary goal of the study is to develop an early (within 4 weeks) combined microbiota/metabolic signature predicting clinical response upon anti-inflammatory treatment in UC patients.

DETAILED DESCRIPTION:
The investigators perform a longitudinal prospective multi-center study for ulcerative colitis (UC) patients with a flare at/and after the time of starting a new treatment and healthy household controls. They will perform intense longitudinal bio-sampling and deep clinical characterization.

With this information the aim is to develop a predictive signature regarding the success of a new ly started anti-inflammatory therapy after an UC flare.

ELIGIBILITY:
Inclusion criteria ulcerative colitis:

1. Signed informed consent
2. Age 18-80 years
3. General ability to understand and follow study procedures, fluency in German, French, or English
4. Diagnosis of ulcerative colitis since ≥3 months
5. Confirmed flare of ulcerative colitis with partial SCCAI score ≥5 points and at least one biomarker supporting intestinal inflammation
6. Planned start with ozanimod, steroids (prednisone ≥20mg/d or equivalent), or a biological (vedolizumab, infliximab, adalimumab, golimumab, ustekinumab)

Exclusion criteria ulcerative colitis

1. Confirmed cytomegalovirus (CMV) reactivation within the previous 2 weeks (tested as part of standard medical practice at the discretion of the responsible physician)
2. C. difficile related diarrhea, or other confirmed infectious diarrhea in the last 4 weeks (tested as part of standard medical practice at the discretion of the responsible physician)
3. Diagnosis of Crohn's disease
4. Current pouch or ileostomy/ colostomy
5. Severe medical, surgical, or psychiatric comorbidities interfering with study procedures

Inclusion criteria controls

1. Signed informed consent
2. Age 18-80 years
3. General ability to understand and follow study procedures, fluency in German, French, or English
4. No current or past diagnosis of inflammatory bowel disease (IBD)
5. No current medical complaints typic for IBD e.g.

   * Diarrhea, severe constipation, abdominal pain, blood in stool, weight loss
   * Slight symptoms (without impact onto daily activities) are permitted
6. No other current relevant gastrointestinal disease or condition plausibly interfering with microbiota assessment according to the discretion of the study physician

Exclusion criteria controls

1. Confirmed cytomegalovirus (CMV) reactivation within the previous 2 weeks
2. C. difficile related diarrhea, or other confirmed infectious diarrhea in the last 4 weeks
3. Diagnosis of Crohn's disease, ulcerative colitis
4. Current pouch or ileostomy/ colostomy
5. Severe medical, surgical, or psychiatric comorbidities interfering with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients/ participants fulfilling inclusion criteria to one of the following groups will be included:
  1. Patients with a flare of ulcerative colitis who meet the inclusion criteria (see above). Inclusion of 120 patients is planned.
  2. Healthy controls. For each patient, a healthy control individual who shares the same living conditions (e.g., spouse or roommate) is attempted. Enrolment of controls will not be enforced but enrolment of ≥100 controls for 120 patients is expected.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Development of a predictive score regarding success of anti-inflammatory therapy after start of a new treatment in ulcerative colitis | 4 months
  The predictive microbiota signature will be developed using machine learning, considering clinical data, microbiota descriptors, and metabolic changes from day 0 to week 4 (see analysis). Clinical response will be defined as a decrease in the simple clinical colitis activity index (SCCAI) score by ≥3 points 25or to a level of ≤2.5 points 26 at 8 weeks after the start of anti-inflammatory treatment.

SECONDARY OUTCOMES:
Predicting clinical remission | 8 weeks
  Assessment of the microbiota/metabolic signature predicting clinical remission (SSCAI <2.5)
Predicting clinical remission | 12 weeks
  Assessment of the microbiota/metabolic signature predicting clinical remission (SSCAI <2.5)
Predicting clinical remission | 6 months
  Assessment of the microbiota/metabolic signature predicting clinical remission (SSCAI <2.5)
Predicting clinical remission | 12 months
  Assessment of the microbiota/metabolic signature predicting clinical remission (SSCAI <2.5)
Predicting calprotectin reduction | 2 weeks
  Assessment of the microbiota/metabolic signature predicting a reduction in fecal calprotectin levels
Predicting calprotectin reduction | 8 weeks
  Assessment of the microbiota/metabolic signature predicting a reduction in fecal calprotectin levels
Predicting calprotectin reduction | 12 weeks
  Assessment of the microbiota/metabolic signature predicting a reduction in fecal calprotectin levels
Predicting calprotectin reduction | 6 months
  Assessment of the microbiota/metabolic signature predicting a reduction in fecal calprotectin levels
Predicting calprotectin reduction | 12 months
  Assessment of the microbiota/metabolic signature predicting a reduction in fecal calprotectin levels
Differential microbiota response to therapy: Ozanimod | 12 months
  Sensitivity analysis in the subgroup treated with Ozanimod in regards to differential signatures in the prediction signature
Differential microbiota response to therapy: TNF-inhibitors | 12 months
  Sensitivity analysis in the subgroup treated with TNF-inhibitors in regards to differential signatures in the prediction signature
Differential microbiota response to therapy: Vedolizumab | 12 months
  Sensitivity analysis in the subgroup treated with Vedolizumab in regards to differential signatures in the prediction signature
Differential microbiota response to therapy: Ustekinumab | 12 months
  Sensitivity analysis in the subgroup treated with Ustekinumab in regards to differential signatures in the prediction signature
Differential microbiota response to therapy: Steroids | 12 months
  Sensitivity analysis in the subgroup treated with Steroids in regards to differential signatures in the prediction signature
Signature differences between ulcerative colitis and healthy controls | 12 months
  Comparison of microbiota/metabolic signatures between ulcerative colitis patients and controls using clustering and differential abundance analysis
Metagenomic substrain assessment | 12 months
  Identification of substrains in patient samples using metagenomic sequencing and follow up their persistence/loss over time
Fatigue assessment | 12 months
  Fatigue severity measured by the fatigue severity scale over time and assessed for reduction after therapy start
Adverse effects | 12 months
  Assessment regarding potential adverse effects in relation medical therapy by screening questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Misselwitz, Prof., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Bern Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Analytic code for generation of the predictive signature will be made available to other researchers
Supporting Information: Analytic Code
Time Frame: With publication of results
Access Criteria: Acess to analytic code will be detailed in the final publication